CLINICAL TRIAL: NCT00303485
Title: A Randomized, Double-blind, Placebo-controlled Study to Determine Time to Onset of Suppression of the Bone Resorption Marker sCTX With Once Monthly Ibandronate in the Treatment of Postmenopausal Osteoporosis
Brief Title: A Study of Bone Turnover Markers in Post-Menopausal Women With Osteoporosis Treated With Monthly Boniva (Ibandronate)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML19334
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-03

CONDITIONS: Post Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Vitamin D; Ibandronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ibandronate (Experimental): Participants received Ibandronate 150 mg tablet once-monthly along with a combination dietary supplement containing vitamin D 200 international units (IU) and elemental calcium 500 mg twice daily with meals for 6 months.
  Interventions: Drug: Vitamin D and calcium supplementation; Drug: ibandronate [Bonviva/Boniva]
- Placebo (Placebo Comparator): Participants received a matching placebo tablet to Ibandronate once-monthly along with a combination dietary supplement containing vitamin D 200 IU and elemental calcium 500 mg twice daily with meals for 6 months.
  Interventions: Drug: Placebo; Drug: Vitamin D and calcium supplementation

INTERVENTIONS:
Drug: Placebo — po monthly for 6 months
  Arms: Placebo
Drug: Vitamin D and calcium supplementation — As prescribed
Drug: ibandronate [Bonviva/Boniva] — 150mg po monthly for 6 months
  Arms: Ibandronate

SUMMARY:
This study will determine the rapidity of suppression of the bone resorption marker sCTX in post-menopausal women with osteoporosis.Other bone turnover markers will also be evaluated. Patients will be randomised to either monthly Boniva 150mg or placebo, in combination with vitamin D and calcium supplementation. The anticipated time on study treatment is approximately 7 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* women who have been newly diagnosed with post-menopausal osteoporosis, requiring treatment;
* naive to bisphosphonate treatment,or had bisphosphonate treatment for a maximum of 3 months, at least 5 years before screening.

Exclusion Criteria:

* patients on hormone replacement therapy (HRT) within the last 3 months;
* patients on other osteoporosis medication within the last 3 months;
* sCTX below lower limit, or above 3 times the upper limit, of normal premenopausal level;
* hypersensitivity to any component of ibandronate;
* contraindication for calcium or vitamin D therapy;
* history of major gastrointestinal upset;
* malignant disease diagnosed within the previous 10 years (except resected basal cell cancer).

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-02; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- United States (7):
  - Beverly Hills, California
  - La Jolla, California
  - Augusta, Georgia
  - Woodbury, Minnesota
  - The Bronx, New York
  - Hopwood, Pennsylvania
  - Madison, Wisconsin
- Puerto Rico (2):
  - Ponce
  - San Juan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 67 participants were enrolled across 9 study centers in the United States. This study was conducted between 06 February 2006 and 21 June 2007. Out of 67 participants enrolled, 66 participants received at least 1 dose of trial medication (49 participants received Ibandronate and 17 participants received placebo).
Period: Overall Study
Arm/Group | Ibandronate | Placebo
Started | 49 | 17
Completed | 48 | 15
Not Completed | 1 | 2
Not completed — Adverse Event/Intercurrent Illness | 0 | 1
Not completed — Failure to return | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Population included all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibandronate | Placebo | Total
Number analyzed (Participants) | 49 | 17 | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (8.64) | 63.0 (8.41) | 64.0 (8.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 17 | 66
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Relative Percent Change in Serum C-terminal Telopeptide of Type 1 Collagen Concentration (sCTX) From Baseline to Day 3
Description: Serum C-terminal Telopeptide of Type 1 Collagen (sCTX) is a biochemical marker for bone turnover that has been shown to detect increased bone resorption, a process by which bone is broken down within the body. It is measured in units of nanograms (ng) per milliliter (mL). The relative change in sCTX was defined as the relative difference between the value at each time point and the value at Baseline, using the following formula: Relative change = (sCTX time point- sCTX Baseline) / (sCTX Baseline) * 100. The sCTX value used for Baseline was the average of the results from the 2 blood samples taken at screening. If 1 of these 2 samples was nonquantifiable or missing, then the Baseline sCTX was the result from the non-missing sample. Baseline visit was defined as Visit 1.
Time Frame: Baseline (Visit 1) and Day 3
Population: This analysis was performed on the ITT Population. The ITT Population included all randomized participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 46 | 16
Percent change | -70.16 [-80.34 to -57.64] | -5.96 [-20.79 to 6.03]
Statistical Analysis 1: Comparison: Ibandronate vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank sum test; Difference in median = -64.20, 95% CI 2-sided [-80.28 to -46.21]

2. Secondary Outcome: Relative Percent Change in Serum C-terminal Telopeptide of Type 1 Collagen (sCTX) Concentration From Baseline Over Time
Description: sCTX is a biochemical marker for bone turnover that has been shown to detect increased bone resorption, a process by which bone is broken down within the body. The relative change in sCTX was defined as the relative difference between the value at each time point and the value at Baseline, using the following formula: Relative change = (sCTX Time point- sCTX Baseline) / (sCTX Baseline) * 100. The sCTX value used for Baseline was the average of the results from the 2 blood samples taken at screening. If 1 of these 2 samples was nonquantifiable or missing, then the Baseline sCTX was the result from the non-missing sample. Baseline visit was defined as Visit 1.
Time Frame: Baseline (Visit 1), Day (D) 3, D7, D14, D21, D28 of Month (M)1, M2, M3, M4, M5, M6
Population: This analysis was performed on the ITT Population. The ITT Population included all randomized participants who received at least 1 dose of study medication. "n" denotes number of participants who received the indicated study drug for each arm.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 47 | 16
Percent change
  M1D1, (n = 46, 16) | -70.16 [-80.34 to -57.64] | -5.96 [-20.79 to 6.03]
  M1D7, (n = 47, 16) | -73.62 [-78.89 to -61.56] | -12.69 [-26.02 to -0.68]
  M1D14, (n = 47, 15) | -61.19 [-74.42 to -51.22] | -21.99 [-28.69 to -8.24]
  M1D21, (n = 46, 16) | -50.98 [-61.39 to -35.94] | -4.46 [-18.73 to 17.69]
  M1D28, (n = 46, 15) | -43.53 [-56.40 to -29.74] | -6.29 [-18.08 to 4.65]
  M2D7, (n = 46, 15) | -75.57 [-80.41 to -66.09] | -7.42 [-19.25 to 14.34]
  M2D14, (n = 45, 16) | -68.51 [-75.19 to -54.20] | -5.01 [-10.92 to 12.12]
  M2D21, (n = 44, 15) | -53.68 [-65.53 to -41.52] | -7.64 [-28.01 to 23.00]
  M2D28, (n = 45, 15) | -50.32 [-60.70 to -44.15] | -14.33 [-25.27 to 14.69]
  M3D7, (n = 44, 15) | -76.58 [-80.25 to -69.94] | -13.84 [-38.85 to 8.88]
  M3D14, (n = 44, 15) | -66.28 [-75.01 to -53.71] | -17.10 [-31.66 to 11.78]
  M3D21, (n = 45, 14) | -59.77 [-65.43 to -39.30] | -21.69 [-38.65 to -0.46]
  M3D28, (n = 46, 16) | -54.49 [-64.04 to -35.16] | -17.13 [-34.36 to 7.12]
  M4D7, (n = 45, 16) | -76.98 [-80.90 to -63.65] | -21.37 [-36.64 to 10.82]
  M4D14, (n = 47, 16) | -69.50 [-76.37 to -57.86] | -6.82 [-26.10 to 11.16]
  M4D21, (n = 45, 15) | -62.80 [-70.48 to -50.71] | -9.97 [-28.34 to 10.49]
  M4D28, (n = 46, 13) | -59.40 [-64.52 to -43.44] | -2.10 [-34.04 to 10.45]
  M5D7, (n = 46, 14) | -75.40 [-80.50 to -67.63] | -2.86 [-41.48 to 10.82]
  M5D14, (n = 44, 14) | -66.08 [-74.65 to -56.06] | -16.42 [-38.26 to 9.82]
  M5D21, (n = 47, 13) | -58.52 [-69.70 to -44.78] | -4.60 [-25.57 to 9.16]
  M5D28, (n = 43, 12) | -54.00 [-63.79 to -43.42] | -31.85 [-42.51 to 3.93]
  M6D7, (n = 45, 12) | -78.09 [-83.84 to -67.97] | -14.59 [-33.11 to 10.87]
  M6D14, (n = 44, 14) | -71.41 [-78.35 to -62.57] | -18.49 [-38.60 to 11.50]
  M6D21, (n = 47, 15) | -67.52 [-72.57 to -58.09] | -15.97 [-49.90 to 19.54]
  M6D28, (n = 46, 15) | -57.97 [-71.74 to -46.84] | -14.92 [-42.56 to 8.47]

3. Secondary Outcome: Relative Percent Change in Bone Specific Alkaline Phosphatase (BSAP) Concentration From Baseline Over Time
Description: BSAP is a biochemical marker of bone formation and measured in units per litre (U/L). The relative percent change in BSAP was defined as the relative difference between the value at each time point and the value at Baseline, using the following formula: Relative change = (BSAP time point- BSAP Baseline) / (BSAP Baseline) * 100. The greater the percent decrease from Baseline, the greater the response to therapy. Baseline visit was defined as Visit 1.
Time Frame: Baseline (Visit 1), Day (D) 7 and D 28 of Month (M)1, M2, M3, M4, M5, M6
Population: This analysis was performed on the ITT Population. The ITT Population included all randomized participants who received at least 1 dose of study medication. 'n' denotes number of participants who received the indicated study drug for each arm.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 47 | 16
Percent change
  M1D7, (n = 47, 16) | 1.30 [-5.92 to 6.64] | -2.42 [-8.14 to 1.60]
  M1D28, (n = 46,15) | -12.24 [-14.45 to -3.19] | -9.78 [-15.85 to -3.38]
  M2D7, (n = 46, 15) | -16.41 [-18.13 to -8.66] | -12.30 [-19.15 to -3.11]
  M2D28, (n = 46,15) | -23.84 [-26.06 to -17.77] | -11.04 [-22.54 to -3.38]
  M3D7, (n = 45, 15) | -22.61 [-30.58 to -21.05] | -12.84 [-25.35 to -6.10]
  M3D28, (n = 45,16) | -29.82 [-34.30 to -26.67] | -13.24 [-26.78 to -1.47]
  M4D7, (n = 44, 16) | -30.26 [-38.05 to -25.15] | -15.64 [-28.44 to -4.89]
  M4D28, (n = 46,14) | -36.88 [-44.16 to -27.78] | -19.71 [-33.17 to -5.74]
  M5D7, (n = 46, 14) | -39.30 [-42.60 to -30.77] | -21.16 [-34.63 to 5.43]
  M5D28, (n = 43,11) | -38.28 [-45.33 to -32.14] | -20.39 [-43.45 to -3.66]
  M6D7, (n = 46, 12) | -38.54 [-44.05 to -33.18] | -13.86 [-42.79 to -8.15]
  M6D28, (n = 47,15) | -40.26 [-45.87 to -25.61] | -19.24 [-37.59 to -5.26]

4. Secondary Outcome: Relative Percent Change in Parathyroid Hormone (PTH) From Baseline to Post Treatment Assessments
Description: Parathyroid hormone (PTH) regulates calcium and phosphate metabolism in bone and kidney, and is measured in picogram/milliliter (pg/mL). The relative percent change in PTH was defined as the relative difference between the value at each time point and the value at Baseline, using the following formula: Relative change = (PTH time point- PTH Baseline) / (PTH Baseline) * 100. Post treatment assessments were done at Baseline, Month (M)1 Day (D)7, and M6D7
Time Frame: Baseline (Visit 1), Month (M)1 Day (D)7, and M6D7
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 49 | 17
Percent change
  Month 1 Day 7 | 37.74 [25.00 to 81.58] | -1.72 [-10.00 to 33.33]
  Month 6 Day 7 | 29.63 [-5.56 to 59.38] | 4.81 [-13.83 to 45.09]

5. Secondary Outcome: Percentage of Participants With a Serum C-terminal Telopeptide of Type1 Collagen (sCTX) Concentration Between 0.011 and 0.631 ng/mL and Who Have Achieved a Decrease in sCTX Concentration of at Least 8 Percent
Description: The Cochran-Mantel Haenszel test stratified by Baseline sCTX category was used to compare the 2 treatment groups for proportion of participants whose sCTX concentration was between 0.011 and 0.631 ng/mL (premenopausal normal range mean +/- 2 SD) who achieved a decrease in sCTX of at least 8% from Baseline. Mean and SD are based on the normal range for premenopausal women: Mean = 0.321 ng/mL, SD=0.155 ng/mL. Baseline visit was defined as Visit 1.
Time Frame: Baseline (Visit 1) and Day (D)3 of Month (M)1 and; D7, D14, D21, D28 of each M1, M2, M3, M4, M5, and M6
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 49 | 17
Percentage of participants
  Baseline, (n = 49, 17) | 59.2 | 58.8
  M1D3, (n = 46,16) | 87.8 | 58.8
  M1D7, (n = 47,16) | 87.8 | 76.5
  M1D14, (n = 47, 15) | 87.8 | 64.7
  M1D21, (n = 46, 16) | 83.7 | 58.8
  M1D28, (n = 46, 15) | 85.7 | 64.7
  M2D7, (n = 46, 15) | 89.8 | 64.7
  M2D14, (n = 45, 16) | 83.7 | 58.8
  M2D21, (n = 44, 15) | 81.6 | 64.7
  M2D28, (n = 45, 15) | 83.7 | 64.7
  M3D7, (n = 44, 15) | 83.7 | 64.7
  M3D14, (n = 44, 15) | 85.7 | 70.6
  M3D21, (n = 45, 14) | 81.6 | 52.9
  M3D28, (n = 46, 16) | 83.7 | 76.5
  M4D7, (n = 45, 16) | 91.8 | 76.5
  M4D14, (n = 47, 16) | 89.8 | 64.7
  M4D21, (n = 45, 15) | 83.7 | 64.7
  M4D28, (n = 46, 13) | 85.7 | 58.8
  M5D7, (n = 46, 14) | 91.8 | 64.7
  M5D14, (n = 44, 14) | 87.8 | 64.7
  M5D21, (n = 47, 13) | 89.8 | 58.8
  M5D28, (n = 43, 12) | 81.6 | 64.7
  M6D7, (n = 45, 12) | 89.8 | 52.9
  M6D14, (n = 44, 14) | 85.7 | 64.7
  M6D21, (n=47, 15) | 91.8 | 64.7
  M6D28, (n = 46,15) | 87.8 | 64.7

6. Secondary Outcome: Percentage of Participants With a Serum C-terminal Telopeptide of Type 1 Collagen (sCTX) Concentration Between 0.011 and 0.476 ng/mL
Description: Percentage of participants whose sCTX concentration was between 0.011 and 0.476 ng/mL (Mean -2 to + 1 SD) were analyzed at particular time points. Mean and SD are based on the normal range for premenopausal women: Mean = 0.321 ng/mL, SD = 0.155 ng/mL. Baseline visit was defined as Visit 1.
Time Frame: Baseline (Visit 1) and Day (D)3 of M1 and D7, D14, D21, D28 of each M1, M2, M3, M4, M5, M6
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 49 | 17
Percentage of participants
  Baseline, (n = 49, 17) | 46.9 | 41.2
  M1D3, (n = 46,16) | 18.4 | 47.1
  M1D7, (n = 47,16) | 10.2 | 58.8
  M1D14, (n = 47, 15) | 24.5 | 47.1
  M1D21, (n = 46, 16) | 22.4 | 47.1
  M1D28, (n = 46, 15) | 32.7 | 52.9
  M2D7, (n = 46, 15) | 8.2 | 52.9
  M2D14, (n = 45, 16) | 14.3 | 52.9
  M2D21, (n = 44, 15) | 24.5 | 58.8
  M2D28, (n = 45, 15) | 30.6 | 64.7
  M3D7, (n = 44, 15) | 14.3 | 52.9
  M3D14, (n = 44, 15) | 16.3 | 47.1
  M3D21, (n = 45, 14) | 20.4 | 35.3
  M3D28, (n = 46, 16) | 26.5 | 52.9
  M4D7, (n = 45, 16) | 14.3 | 64.7
  M4D14, (n = 47, 16) | 14.3 | 47.1
  M4D21, (n = 45, 15) | 18.4 | 41.2
  M4D28, (n = 46, 13) | 22.4 | 41.2
  M5D7, (n = 46, 14) | 10.2 | 41.2
  M5D14, (n = 44, 14) | 18.4 | 47.1
  M5D21, (n = 47, 13) | 20.4 | 41.2
  M5D28, (n = 43, 12) | 20.4 | 41.2
  M6D7, (n = 45, 12) | 8.2 | 29.4
  M6D14, (n = 44, 14) | 12.2 | 47.1
  M6D21, (n=47, 15) | 22.4 | 35.3
  M6D28, (n = 46, 15) | 18.4 | 47.1

7. Secondary Outcome: Percentage of Participants With a Serum C-terminal Telopeptide of Type 1 Collagen (sCTX) Concentration Between 0.011 and 0.321 ng/mL
Description: Percentage of participants whose sCTX concentration was between 0.011 and 0.321 ng/mL (Mean -2 to + 0 SD) were analyzed at particular time points. Mean and SD are based on the normal range for premenopausal women: Mean = 0.321 ng/mL, SD = 0.155 ng/mL.
Time Frame: Baseline (Visit 1), Day (D)3 of M1, and D7, D14, D21, D28 of each M1, M2, M3, M4, M5, M6
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 49 | 17
Percentage of participants
  Baseline, (n = 49, 17) | 16.3 | 23.5
  M1D3, (n = 46,16) | 6.1 | 29.4
  M1D7, (n = 47,16) | 2.0 | 35.3
  M1D14, (n = 47, 15) | 8.2 | 11.8
  M1D21, (n = 46, 16) | 10.2 | 17.6
  M1D28, (n = 46, 15) | 18.4 | 23.5
  M2D7, (n = 46, 15) | 6.1 | 23.5
  M2D14, (n = 45, 16) | 6.1 | 29.4
  M2D21, (n = 44, 15) | 8.2 | 35.3
  M2D28, (n = 45, 15) | 6.1 | 29.4
  M3D7, (n = 44, 15) | 4.1 | 23.5
  M3D14, (n = 44, 15) | 4.1 | 35.3
  M3D21, (n = 45, 14) | 8.2 | 17.6
  M3D28, (n = 46, 16) | 4.1 | 23.5
  M4D7, (n = 45, 16) | 4.1 | 29.4
  M4D14, (n = 47, 16) | 2.0 | 17.6
  M4D21, (n = 45, 15) | 0.0 | 17.6
  M4D28, (n = 46, 13) | 6.1 | 11.8
  M5D7, (n = 46, 14) | 2.0 | 11.8
  M5D14, (n = 44, 14) | 4.1 | 23.5
  M5D21, (n = 47, 13) | 6.1 | 17.6
  M5D28, (n = 43, 12) | 8.2 | 17.6
  M6D7, (n = 45, 12) | 4.1 | 17.6
  M6D14, (n = 44, 14) | 4.1 | 23.5
  M6D21, (n= 47, 15) | 10.2 | 23.5
  M6D28, (n = 46,15) | 6.1 | 29.4

8. Secondary Outcome: Difference Between the Minimum and Maximum Relative Percent Change in Serum C-terminal Telopeptide of Type 1 Collagen (sCTX) Concentrations
Description: Overall minimum and maximum relative percent change in sCTX concentrations from Baseline were calculated for all participants over D7, D14, D21 and D28 of Month 6 and the difference between it was analyzed.
Time Frame: Day (D)7, D14, D21 and D28 of Month 6
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 48 | 15
Percent change | 17.23 [1.7 to 55.9] | 22.89 [11.3 to 44.1]

9. Secondary Outcome: Number of Participants With Any Marked Abnormality in Laboratory Parameters
Description: Marked laboratory abnormalities are those which exceed the marked abnormality range (i.e., greater or less than the Roche defined marked abnormality range; i.e Low or High) and which also represents a clinically relevant change from Baseline of at least a designated amount. The indicated abnormal laboratory parameters (along with their marked reference range) are as follows : Hematocrit (0.31- 0.56 fraction), hemoglobin (110 - 200 g/L), platelets (100 - 550 *10^9/L), white blood cell (WBC) (3.0 - 18.0 *10^9/L), alanine aminotransferase (ALT) (0 - 110 U/L), creatinine (0 - 154 µmol/L), chloride (95 - 115 mmol/L), phosphate (0.75 - 1.60 mmol/L ). Creatinine clearance was calculated using the Cockroft-Gault formula.
Time Frame: Up to 7 months
Population: The Safety analysis Population was a subset of the ITT Population consisting of participants with at least 1 post-baseline safety assessment. 'n' denotes the number of participants who received the indicated study drug for each arm.
Measure: Number; unit: Participants
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 48 | 16
Participants
  Hematocrit-Low, (n = 46,16) | 1 | 0
  Hemoglobin-Low, (n = 46, 16) | 1 | 0
  Platelets-High, (n = 46, 15) | 0 | 1
  White blood cells-Low, (n = 46, 16) | 2 | 0
  ALT- High, (n = 48, 16) | 1 | 0
  Creatinine-High, (n = 48, 16) | 1 | 0
  Chloride-Low, (n = 48, 16) | 0 | 1
  Potassium-High, (n = 48, 16) | 0 | 1
  Phosphate-High, (n = 48, 16) | 1 | 0

10. Secondary Outcome: Number of Participants With Any Adverse Event or Serious Adverse Event
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. A Serious Adverse Event (SAE) is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect.
Time Frame: Up to 7 months
Population: The Safety Analysis Population was a subset of the ITT Population consisting of participants with at least 1 post-baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | Ibandronate | Placebo
Number analyzed (Participants) | 49 | 17
Participants
  Any AEs | 40 | 12
  Any SAEs | 1 | 2

ADVERSE EVENTS:
Time Frame: Up to 7 months
Description: Serious adverse events (SAEs) and non-serious AEs were reported for members of the safety population which included all enrolled participants who had received at least one dose of study medication and who had at least one post-baseline safety follow-up assessment.
Arm/Group | Ibandronate | Placebo
Serious Adverse Events (participants affected / at risk) | 1/49 | 2/17
Other Adverse Events (participants affected / at risk) | 28/49 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate (N=49) | Placebo (N=17)
Angina Unstable (Cardiac disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate (N=49) | Placebo (N=17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Nasopharyngitis (Infections and infestations) | 8 | 5
Diarrhoea (Gastrointestinal disorders) | 7 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Headache (Nervous system disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.